CLINICAL TRIAL: NCT03883061
Title: Mathematical Modeling and Risk Factor Analysis for Mortality of Sepsis Based on Real World Data in China
Brief Title: Mathematical Modeling and Risk Factor Analysis for Mortality of Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: Department of Emergence, The First Hospital Affiliated to South China University, Hengyang, Hunan, China. (Unknown); Department of Integrative Medicine, Huashan Hospital of Fudan University, Shanghai, China (Unknown); Department of Biomedical Informatics and Statistics, Insitute of Integrative Medicine, Fudan University, Shanghai, China (Unknown); Department of emergence, Hunan people's hospital, Changhai, Hunan, China (Unknown); Department of emergence, The hospital affiliated to Jining medical college, Jining, Shandong, China (Unknown); Department of emergence, Huaihua people's hospital, Huaihua, Hunan, China (Unknown)
Responsible Party: Principal Investigator, Zihui Tang, Associate Professor, Huashan Hospital
Other Study IDs: 20190319
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Morality; Risk Factor, Sepsis; Predictive Model
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mortality of sepsis: the study sample would be extracted from electronic health records in emergence departments. risk factor analysis and mathematical modeling would be performed to evaluate the significant and independent risk factors and predictive models.
  Interventions: Other: regular medical treatment

INTERVENTIONS:
Other: regular medical treatment — regular medical treatment

SUMMARY:
The purpose of this study was to investigate the risk factors for mortality of sepsis and to create mathematical models to predict the survival rate based on electronic health records that extracted from hospital information system. More than 1000 records should be collected and used to data analysis. Univariate and multivariable logistic regression model were applied to risk factors analysis for the outcome, and machine learn algorithms were employed to generate predictive models for the outcome.

ELIGIBILITY:
Inclusion Criteria:

* all records with sepsis in emergence department of hospitals

Exclusion Criteria:

* subjects with major missing data

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with sepsis in emergence department of hospitals
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality of sepsis | 4 weeks
  mortality of sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- Zihui Tang, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu Y, Tang ZH, Zeng F, Li Y, Zhou L. The association and predictive value analysis of metabolic syndrome combined with resting heart rate on cardiovascular autonomic neuropathy in the general Chinese population. Diabetol Metab Syndr. 2013 Nov 17;5(1):73. doi: 10.1186/1758-5996-5-73. PMID 24238358